CLINICAL TRIAL: NCT03830879
Title: Shenzhen Birth Cohort Study
Status: Recruiting | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Li Cai, Associate professor, Sun Yat-sen University
Other Study IDs: SZBCS
Record Dates: First submitted 2019-01-30; First posted 2019-02-05 (Actual); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Pregnancy Complications; Gestational Diabetes; Obstetric Labor Complications; Neurodevelopmental Disorders; Childhood Obesity
MeSH Terms: conditions — Pregnancy Complications; Diabetes, Gestational; Obstetric Labor Complications; Neurodevelopmental Disorders; Pediatric Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — During pregnancy: maternal blood, urine, hair and toenails. At delivery: umbilical cord blood, placenta , umbilical cord, meconium, mother's saliva and milk. During infancy: dry blood spot, stool and blood. During childhood: Mother's saliva, milk, baby's saliva and feces.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- No treatment: This cohort study have any no treatment.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This cohort study have any no intervention.

SUMMARY:
The Shenzhen Birth Cohort Study was set up to investigate the effect of early life environmental exposures on short- and long-term health consequences in Shenzhen, China.

DETAILED DESCRIPTION:
Shenzhen Birth Cohort (Xinmiao Project) is a scientific research/public health project under the support of Shenzhen city and Nanshan district, which was jointly initiated by Nanshan Maternity and Child Healthcare Hospital of Shenzhen and school of public health, Sun Yat-sen University. The project plans to recruit 10,000 participants in early pregnancy and follow up for seven years in the first stage. Biological samples, questionnaires and data for child growth and development, disease and health will be collected. The study is aimed to provide evidence for DOHaD Hypothesis and find the prevention and control measures for some childhood diseases. The core members of the research team are composed of experts from different disciplines in the field of public health, including 4 professors and 3 associate professors. With the support of an executive sponsor, the project is undertaken by the Birth Cohort Study Center. Currently, the center has 3 staff form hospital (one doctor and two masters ) and 5-7 master candidates from Sun Yat-sen University. It is an energetic and enthusiastic team.

ELIGIBILITY:
Inclusion Criteria:

* 1. Pregnant women plan to delivery and participate in child care in our hospital; 2. Pregnant women plan to reside in Shenzhen for at least 7 years; 3. Pregnant women who show interest in the study and agree to provide informed consent; 4. Gestational weeks are less than 20 weeks.Those who will agree that their neonatal will be included in the study and be followed up regularly in our child health clinic until an age of 7 years.

Exclusion Criteria:

* Pregnant women who have been pregnant for more than 20 weeks; refuse to participate; unable to guarantee delivery in our hospital or can't participate in child care in our hospital; mentally incapacitated and need guardians; or be unwilling to sign informed consent.

Ages: 15 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Pregnant women attending their first routine antenatal examinations and their partners and offspring.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2018-03-06 (Actual); Primary Completion 2025-03-05 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Fetal outcomes. | At delivery.
  Including intrauterine growth retardation, abortion, stillbirth, live birth, preterm. birth, low birth weight, macrosomia and birth defects.

SECONDARY OUTCOMES:
Maternal weight changes (kg). | At pre-pregnancy period, 20 weeks of gestation, 28 weeks of gestation, the time before labor and 30 days after delivery.
  Assess using electronic weighing machine.
Number of participant with gestational complications. | At delivery.
  Including gestational hypertension and preeclampsia, and gestational diabetes mellitus.
Number of participant with postnatal depression. | At 30 days after delivery, 3 months, 6 months after delivery.
  Assess using Edinburgh Postnatal Depression Scale (EPDS).
Physical development. | at age of 1 month, 3 months, 6months, 1 year, 3 years and 6 years.
  Including weight changes (kg) and height changes (cm).
Neurodevelopment. | at age of 1 month, 3 months, 6months, 1 year, 3 years and 5 years.
  Including gross motor, fine motor, language, and social function, assess using Ages and Stages Questionnaires (ASQ-3 and ASQ-SE).

CONTACTS AND LOCATIONS:
Locations (1):
- RuiGao, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided